## **Cover Page**

## **Consent Form**

Study Title: Taste Perception, Salivary Proteins, & the Oral Microbiome

Document Date: 08/08/2022

NCT Number: NCT04107688

| ID# |
|-----|
|-----|

## **CONSENT FORM**

## Study on Astringency Perception: Individual Differences and Salivary Mechanisms Taste Perception, Astringency and the Oral Microbiome

Principal Investigator: Beverly J. Tepper, Ph.D.

Sensory Evaluation Laboratory (Room 211)
Department of Food Science, Rutgers University
65 Dudley Road, New Brunswick, NJ 08901
848-932-5417 Email: <a href="mailto:btepper@sebs.rutgers.edu">btepper@sebs.rutgers.edu</a>

**PURPOSE:** Genetic differences in taste are believed to play an important role in food selection, especially for strong-tasting foods and beverages. The overall goal of this project is to better understand how genes that control food preferences differ among people and whether saliva composition and oral health is related to these differences. You are invited to participate in this research because you have already participated in a screening procedure and you qualify for this study.

**PROCEDURES:** You will be asked to participate in a 2-week study. During days 1-3, you will rinse your mouth with plain water in the morning and evening each day as part of your normal daily routine. During days 4-14, you will rinse with a cranberry-derived oral rinse twice a day. This oral rinse will be provided to you along with the proper instructions on using it. You will come to the lab for two test sessions; one on day 3 and one on day 14. During the two sessions, you will be asked to evaluate food samples as well as provide saliva samples by spitting into a plastic tube. Each session will take approximately 30 minutes to complete. The saliva samples will be analyzed for salivary protein profiles and microbial profiles (oral microbiome). The study activities and timeline is attached.

**RISKS:** Use of the cranberry-derived rinse and the saliva collection procedure poses no foreseeable risks to your health.

**BENEFITS:** Although you will receive no direct benefits from participating in this study, this research will benefit society by providing a better understanding of the relationship between taste and oral health.

**COMPENSATION:** At the completion of the study, you will receive a single payment of \$ 50.

**CONFIDENTIALITY:** The information collected in this screening will be kept strictly confidential. 'Confidential' means that your name and the information collected about you will be linked by a code number, and the code number will be used to identify your data. All data will be kept in a locked filing cabinet or on a pass-word protected computer in the Principal Investigator's laboratory. Only research staff involved in this study or the Institutional Review Board (a committee that reviews research studies in order to protect research participants) at Rutgers University will be allowed to see the data, except as may be required by law. If a report of this study is published, or the results are presented at a professional conference, only group results will be stated. You will not be personally identified in any report of this research.

**YOUR RIGHTS AS A RESEARCH PARTICIPANT:** Your participation in this study is completely voluntary and you have the right to withdraw at any time without explanation or penalty.

**DISCLAIMER:** Rutgers University has made no general provision for financial compensation or medical treatment for any physical injury resulting from this research.

| Initials | Pg | 1 | of | 2 | • |
|----------|----|---|----|---|---|
|----------|----|---|----|---|---|

**CONTACT INFORMATION:** You can contact the Principal Investigator at the number listed above if you have any questions about this study.

If you have any questions about your rights as a research subject, you may contact the IRB Administrator at Rutgers University at:

Arts and Sciences Institutional Review Board for the Protection of Human Subjects Office of Research and Regulatory Affairs
Rutgers University, the State University of New Jersey
335 George Street
Liberty Plaza / 3rd Floor / Suite 3200

New Brunswick, NJ 08901

| Tel: 732-235-2866 | Email: | human-sub | jects@ | ored.rut | gers.edu |
|-------------------|--------|-----------|--------|----------|----------|
|-------------------|--------|-----------|--------|----------|----------|

| Name of participant (print) | Date |
|---|---|
| Signature of Participant | Signature of Investigator |
| Please confirm that you received a copy of this st | tatement for your records (initials) |

This informed consent form was approved by the Rutgers Institutional Review Board for the Protection of Human Subjects on \_\_\_\_\_; approval of this form expires on \_\_\_\_\_